CLINICAL TRIAL: NCT04323696
Title: Comparison of Staple Line Suturing Reinforcement Methods in Laparoscopic Sleeve Gastrectomy
Brief Title: Comparison of Staple Line Suturing in Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Zubaidah Nor hanipah, Associate Professor Dr, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 53293
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: All patients who underwent laparoscopic sleeve gastrectomy from March 2020 till February 2021 will be included
Who Masked: Participant
Masking Description: This is a single blinded randomisation whereby the patient is not aware on the staple-line suturing reinforcement used. Suturing reinforcement of the staple-line is our standard of care in all laparoscopic sleeve gastrectomy patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Over-sewing (Other): Patients under over-sewing arm are subjected to staple line reinforcement using over-sewing method
  Interventions: Procedure: Staple line suturing reinforcement methods - Plication and Over-sewing
- Plication (Other): Patients under over-sewing arm are subjected to staple line reinforcement using plication method
  Interventions: Procedure: Staple line suturing reinforcement methods - Plication and Over-sewing

INTERVENTIONS:
Procedure: Staple line suturing reinforcement methods - Plication and Over-sewing — Sleeve gastrectomy procedure will be performed laparoscopically. The greater curvature of the stomach will be mobilised, and stomach will be sleeved using 39F calibration tube as the stent using 5-6 60 mm-stapler reloads depending on the length and thickness of the stomach. The staple-line is then reinforced using 3/0 absorbable sutures continuously throughout the staple-line. The two staple-line suturing methods in this study include over-sewing (through and through) and plication (Lembert).

SUMMARY:
Sleeve gastrectomy (SG) involves the creation of small gastric reservoir based on lesser curvature of the stomach, which is fashioned by a longitudinal gastrectomy that preserves the antrum and pylorus together with its vagal innervation. Recently SG is viewed as a multi-purpose bariatric procedure that restricts the stomach size to induce satiety and resects fundal ghrelin-producing cells to decrease appetite. However, the risk of staple line leak and bleeding remains one of its challenging complications. Despite the fact that there are a large number of studies assessing various methods of making the staple line secure, there is to date, no consensus on which technique is best for reducing the risk of stapler line bleeding and leak. Hence, this study aims to compare staple line suturing reinforcement methods in sleeve gastrectomy using plication and over-sewing techniques.

ELIGIBILITY:
Inclusion Criteria:

- Patients at our Bariatric Clinic fulfilling NIH criteria for bariatric surgery and planned operation of laparoscopic sleeve gastrectomy as primary bariatric procedure will be evaluated for possible inclusion

Exclusion Criteria:

1. Age < 18 or > 65
2. BMI < 35 and > 60 kg/m2
3. American Society of Anesthesiologists (ASA) score > 3
4. Concurrent surgical procedure including:

   1. ventral hernia repair
   2. cholecystectomy
   3. hiatal hernia repair with posterior cruroplasty
   4. extensive lysis of adhesions
   5. other procedures that mandate addition of 'trocar(s)' or 'feeding tube'

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Immediate and early post-operative complication | 0-30 days
  Staple line bleeding

SECONDARY OUTCOMES:
Immediate and early post-operative complication | 0-30 days
  Staple line leak
Immediate and early post-operative complication | 0-30 days
  Re-admission and re-operation